CLINICAL TRIAL: NCT07287566
Title: The Impact of Different Methods of Oral Hygiene on Incidence of Ventilator Associated Pneumonia in Pediatric Intensive Care Unit
Brief Title: Impact of Oral Care on Ventilator Associated Pneumonia
Acronym: OH-VAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU MS407 /2024; FMA MS407 /2024 (Other: Research Ethics Committee-Faculty of Medicine-ASU)
Record Dates: First submitted 2025-11-20; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Ventilator Associated Pneumonia ( VAP)
Keywords: oral hygiene; ventilator associated pneumonia; chlorohexidine; mechanical ventilation; pediatric intensive care unit
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Toothbrushing; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): Toothbrushing + Chlorohexidine
  Interventions: Procedure: Toothbrushing + Chlorhexidine
- control group (Active Comparator): Routine oral care + Chlorohexidine
  Interventions: Procedure: Routine oral care + Chlorohexidine

INTERVENTIONS:
Procedure: Toothbrushing + Chlorhexidine — three times daily for 5 minutes
  Arms: intervention group
Procedure: Routine oral care + Chlorohexidine — three times daily for 5 minutes
  Arms: control group

SUMMARY:
The goal of this clinical trial was to find out whether cleaning the mouths of children in the Pediatric Intensive Care Unit (PICU) with toothbrushing and chlorhexidine lowers the chance of getting lung infections in patients on breathing machines compared to routine mouth care. The study determined whether this approach changed how long children need a breathing machine, how many days they stayed in the PICU, and whether it affects survival. The main questions it aimed to answer were:

* Did toothbrushing with chlorhexidine, compared to routine mouth care, lowered the risk of lung infections in patients on breathing machines in the PICU?
* Did this approach also affect recovery outcomes, including duration of needing a breathing machine, length of PICU stay, and survival rates?

Researchers compared toothbrushing and chlorhexidine to routine mouth care to see if toothbrushing and chlorhexidine lowered the risk of lung infections in patients on breathing machines.

Participants:

Had safety practices to prevent lung infections in patients on breathing machines Had toothbrushing and chlorhexidine or routine mouth care three times daily 5 minutes in each Had physical check-up and any tests needed as part of their care

DETAILED DESCRIPTION:
Pediatric dentist trained the nurses to follow the proper oral care protocol. Safe practices as keeping the patient's head slightly raised while lying in bed and clean the patients mouth regularly to remove germs. Participants and researcher didn't know which oral care method was being administered making this double blinded study. The participants were divided into two groups 59 patients in each group. In Tooth brushing group, tooth paste and soft tooth brush was positioned at 45 degree angle with a firm gentle pressure, brushing back and forth or using a circular motion 15 to 20 times before moving to the next area for one minute plus application of chlorhexidine mouthwash to a swab on the oral mucosa, teeth, gums, hard palate, and tongue, followed by 20 milliliter (mL) of normal saline, the procedure was finished with hypo pharyngeal suctioning. In routine oral care group only a swab with chlorhexidine and rubbing it on the surface of the tongue, gum and mucosa followed by 20 mL of normal saline, the procedure was finished with hypo pharyngeal suctioning.

investigations include laboratory (Complete blood picture, C-reactive protein and Venous blood gases (VBG) were done. Radiological and microbiological included sputum culture collected on fifth day were also done.

ELIGIBILITY:
Inclusion Criteria: dentate mechanically ventilated

-

Exclusion Criteria:

* primary immune deficiency coagulation disorders jaw fractures

Ages: 18 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
incidence of VAP in pediatric patients in PICU receiving toothbrushing and chlorohexidine in comparison to routine oral hygiene | Baseline, Day 2, Day3, Day 4 and Day 5 of enrollment
  number of patients who develop VAP

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed R. Ahmed, MD, Principal Investigator — Ain Shams University
Locations (1):
- Pediatric Intensive Care Units, Children Hospital, Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
no plan to share

REFERENCES:
- [Result] de Lacerda Vidal CF, Vidal AK, Monteiro JG Jr, Cavalcanti A, Henriques APC, Oliveira M, Godoy M, Coutinho M, Sobral PD, Vilela CA, Gomes B, Leandro MA, Montarroyos U, Ximenes RA, Lacerda HR. Impact of oral hygiene involving toothbrushing versus chlorhexidine in the prevention of ventilator-associated pneumonia: a randomized study. BMC Infect Dis. 2017 Jan 31;17(1):112. doi: 10.1186/s12879-017-2188-0. PMID 28143414
- See also: The Egyptian Journal of Critical Care Medicine. 5(3):87-91. — https://doi.org/10.1016/j.ejccm.2017.11.002
- See also: Prevention of VAP: Endless evolving evidences-systematic literature review. — https://pubmed.ncbi.nlm.nih.gov/34091899/

DOCUMENTS (2):
  • Study Protocol (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT07287566/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT07287566/SAP_001.pdf